CLINICAL TRIAL: NCT01164579
Title: An Exploratory Phase 2, Randomized, Double-blind, Multicenter Study To Assess The Effects Of Tofacitinib (Cp-690,550) On Magnetic Resonance Imaging Endpoints, In Methotrexate Naive Subjects With Early Active Rheumatoid Arthritis
Brief Title: Effects of Tofacitinib (CP-690,550) on Magnetic Resonance Imaging (MRI)- Assessed Joint Structure In Early Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921068; 2010-020890-18 (EudraCT Number)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis; Joint Structure; Magnetic Resonance Imaging; Janus Kinase (JAK) Inhibitor; Tasocitinib; Tofacitinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tofacitinib (CP 690,550) 10 mg BID plus MTX (Experimental)
  Interventions: Drug: Tasocitinib plus Methotrexate
- Tofacitinib (CP-690,550) 10 mg BID, tablet plus placebo MTX (Experimental)
  Interventions: Drug: Tofacitinib plus placebo methotrexate
- Placebo tofacitinib (CP-690,55) plus MTX 10 mg/wk to 20 mg/wk (Active Comparator)
  Interventions: Drug: Placebo tofacitinib plus Methotrexate

INTERVENTIONS:
Drug: Tasocitinib plus Methotrexate — Tofacitinib (CP 690,550) 10 mg BID, tablets + methotrexate (MTX) 10 mg/wk to 20 mg/wk, titrated over 2 months
  Arms: Tofacitinib (CP 690,550) 10 mg BID plus MTX
Drug: Tofacitinib plus placebo methotrexate — Tofacitinib (CP-90,550) 10 mg BID, tablets. Placebo to match methotrexate (MTX) capsules titrated as in Treatment Arm 1.
  Arms: Tofacitinib (CP-690,550) 10 mg BID, tablet plus placebo MTX
Drug: Placebo tofacitinib plus Methotrexate — Methotrexate (MTX) 10 mg/wk to 20 mg/wk, capsules, titrated over 2 months. Placebo in tablets to match tofacitinib
  Arms: Placebo tofacitinib (CP-690,55) plus MTX 10 mg/wk to 20 mg/wk

SUMMARY:
Evaluation of efficacy and safety of tofacitinib (CP-690,550) for the treatment of early rheumatoid arthritis in adult patients with moderate to severe disease who are methotrexate naïve. The efficacy will be evaluated by exploring the effects on joint structure assessed by magnetic resonance imaging, x-rays and by standard clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with moderate to severe early rheumatoid arthritis (< 2 years) who are methotrexate and biologic disease modifying antirheumatic drug naive.

Exclusion Criteria:

* Pregnant or lactating patients;
* Patients with renal or hepatic impairment or other severe or progressing disease;
* Patients with contraindication to magnetic resonance imaging with gadolinium contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (8):
  - ArthroCare, Arthritis Care & Research, PC, Gilbert, Arizona
  - Talbert Medical Group, Huntington Beach, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Millennium Research, Ormond Beach, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - St. Petersburg Arthritis Center, St. Petersburg, Florida
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Office of John P. Lavery, MD, PA, Allen, Texas
- Argentina (3):
  - OMI - Organización Médica de Investigación, Buenos Aires
  - Saint Dennis Medical Group S.A., Buenos Aires
  - Consultorios Reumatologicos Pampa, Buenos Aires
- Chile (2):
  - Consulta Privada Dr. Juan Ignacio Vargas, Osorno, Los Lagos Region
  - Hospital Base Valdivia, Valdivia, Region XIV
- Croatia (2):
  - University Hospital Centre Split,Department for Internal Medicine, Division of Clinical Rheumatology, Split
  - General Hospital Sveti Duh, Zagreb
- Czechia (8):
  - ARTMEDI UPD s r.o., Hostivice
  - Nemocnice na Frantisku s poliklinikou, Prague
  - Nemocnice na Frantisku, Prague
  - Revmatologicky ustav, Prague
  - DC Mediscan, Praha 11 - Chodov
  - Uherskohradistska nemocnice, a.s., Uherské Hradiště
  - Nemocnice Atlas, a.s., Zlín
  - PV-Medical s.r.o., Zlín
- Hungary (5):
  - Drug Research Center Kft., Balatonfüred
  - Orszagos Reumatologiai es Fizioterapias Intezet, Budapest
  - Synexus Magyarorszag Kft., Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Reumatologiai Tanszek, Debrecen
  - Petz Aladar Megyei Oktato Korhaz/Reumatologiai es Mozgasszervi Rehabilitacios Centrum, Győr
- Mexico (7):
  - Centro de Investigacion y Tratamiento Reumatologico S.C., México, D. F.
  - Hospital Angeles Mocel, México, D.f.
  - Centro de Investigacion y Tratamiento Reumatologico SC, Mexico City, Mexico City
  - Hospital Angeles Mocel, Mexico City, Mexico City
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi S.C., San Luis Potosí City, San Luis Potosí
  - Hospital Angeles Mocel, Chapultepec
  - Investigacion y Biomedicina de Chihuahua S.C, Chihuahua City
- Poland (3):
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Osteoporozy i Chorob Kostno-Stawowych J., Bialystok
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj, Poznan
  - Nzoz "Nasz Lekarz", Torun
- Puerto Rico (2):
  - Mindful Medical Research, San Juan, PR
  - San Juan Arthritis & Research Center, San Juan

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] van der Heijde D, Landewe RBM, Wollenhaupt J, Strengholt S, Terry K, Kwok K, Wang L, Cohen S. Assessment of radiographic progression in patients with rheumatoid arthritis treated with tofacitinib in long-term studies. Rheumatology (Oxford). 2021 Apr 6;60(4):1708-1716. doi: 10.1093/rheumatology/keaa476. PMID 33057725
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Conaghan PG, Ostergaard M, Troum O, Bowes MA, Guillard G, Wilkinson B, Xie Z, Andrews J, Stein A, Chapman D, Koenig A. Very early MRI responses to therapy as a predictor of later radiographic progression in early rheumatoid arthritis. Arthritis Res Ther. 2019 Oct 21;21(1):214. doi: 10.1186/s13075-019-2000-1. PMID 31639034
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Conaghan PG, Ostergaard M, Bowes MA, Wu C, Fuerst T, van der Heijde D, Irazoque-Palazuelos F, Soto-Raices O, Hrycaj P, Xie Z, Zhang R, Wyman BT, Bradley JD, Soma K, Wilkinson B. Comparing the effects of tofacitinib, methotrexate and the combination, on bone marrow oedema, synovitis and bone erosion in methotrexate-naive, early active rheumatoid arthritis: results of an exploratory randomised MRI study incorporating semiquantitative and quantitative techniques. Ann Rheum Dis. 2016 Jun;75(6):1024-33. doi: 10.1136/annrheumdis-2015-208267. Epub 2016 Jan 25. PMID 27002108
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921068&StudyName=Effects%20of%20Tofacitinib%20%28CP-690%2C550%29%20on%20Magnetic%20Resonance%20Imaging%20%28MRI%29-%20Assessed%20Joint%20Structure%20In%20Early%20Rheumatoid%20Arthritis%20%28R

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib (CP-690,550) Plus Methotrexate (MTX): Participants received CP-690,550 10 milligrams (mg), tablets, orally (PO), twice daily (BID), and MTX 10 mg per week (mg/week) to 20 mg/week, capsules, PO, for a maximum of 12 months. MTX dose was titrated as follows: 10 mg once weekly for 4 weeks; if well tolerated, then at Month 1 titrate up to 15 mg once weekly for 4 weeks; if well tolerated, then at Month 2 titrate up to 20 mg once weekly for the duration of the study. A single dose reduction of MTX 5 mg was allowed because of lack of tolerance, as long as the participant remained on a dose of at least MTX 10 mg weekly. Participants also received folate supplementation according to local MTX label guidelines and standard of care.
- Tofacitinib (CP-690,550): Participants received CP-690,550 10 mg tablets, PO, BID and matching placebo MTX capsules, PO, once weekly for a maximum of 12 months. To maintain the blind, matching placebo MTX was titrated as follows: 4 capsules once weekly for 4 weeks; if well tolerated, at Month 1 titrate up to 6 capsules once weekly for 4 weeks; if well tolerated, then at Month 2 titrate up to 8 capsules once weekly for the duration of the study. A single dose reduction of MTX placebo to 2 capsules was allowed because of lack of tolerance, as long as the participant remained on a dose of at least 4 MTX placebo capsules weekly. Participants also received folate supplementation according to local MTX label guidelines and standard of care.
- Methotrexate: Participants received MTX 10 mg/week to 20 mg/week, capsules, PO, and matching placebo CP-690,550 tablets, PO, BID. MTX dose was titrated as follows: 10 mg once weekly for 4 weeks; if well tolerated, then at Month 1 titrate up to 15 mg once weekly for 4 weeks; if well tolerated, then at Month 2 titrate up to 20 mg once weekly for the duration of the study. A single dose reduction of MTX 5 mg was allowed because of lack of tolerance, as long as the participant remained on a dose of at least MTX 10 mg weekly. Participants also received folate supplementation according to local MTX label guidelines and standard of care.
Period: Overall Study
Arm/Group | Tofacitinib (CP-690,550) Plus Methotrexate (MTX) | Tofacitinib (CP-690,550) | Methotrexate
Started | 36 | 36 | 37
Completed | 28 | 27 | 21
Not Completed | 8 | 9 | 16
Not completed — Lack of Efficacy | 0 | 0 | 6
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 3
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Adverse Event | 4 | 2 | 5
Not completed — Reason not specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who were randomized to study medication and received at least 1 dose of randomized study medication.
Groups:
- Tofacitinib (CP-690,550) Plus MTX: Participants received CP-690,550 10 mg, tablets, PO, BID, and MTX 10 mg/week to 20 mg/week, capsules, PO, for a maximum of 12 months. MTX dose was titrated as follows: 10 mg once weekly for 4 weeks; if well tolerated, then at Month 1 titrate up to 15 mg once weekly for 4 weeks; if well tolerated, then at Month 2 titrate up to 20 mg once weekly for the duration of the study. A single dose reduction of MTX 5 mg was allowed because of lack of tolerance, as long as the participant remained on a dose of at least MTX 10 mg weekly. Participants also received folate supplementation according to local MTX label guidelines and standard of care.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate | Total
Number analyzed (Participants) | 36 | 36 | 37 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.3) | 50.8 (12.8) | 47.8 (11.6) | 48.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 29 | 90
  Male | 5 | 6 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 3 in Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS) Wrist and Metacarpophalangeal (MCP) Synovitis
Description: Synovitis is defined as an area in the synovial compartment that shows above normal postgadolinium enhancement of a thickness greater than the width of the normal synovium. T1-weighted images were acquired before and after the administration of intravenous contrast agent containing gadolinium. Intravenous contrast was required to demonstrate enhancing synovitis. Synovitis was scored 0 to 3 in 3 wrist regions and in each of the first through fifth MCP joints. A score of 0 is normal, with no enhancement or enhancement up to the thickness of normal synovium, while scores of 1 to 3 (mild, moderate, severe) refer to increments of one-third of the presumed maximum volume of enhancing tissue in the synovial compartment. Total synovitis score ranges from a minimum of 0 to a maximum of 24. A negative value in synovitis change from Baseline score indicates an improvement.
Time Frame: Month 3
Population: Evaluable Set: all randomized participants who received at least 1 dose of the randomized investigational drug and for whom a variable is nonmissing at both baseline and the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 30 | 32 | 31
score on a scale | -0.80 (0.41) | -0.69 (0.40) | -0.17 (0.40)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Test type: Superiority or Other; p = 0.2696, mixed model repeated measures analysis — 2-sided p-value; alpha equals (=) 0.10; Difference in least squares (LS) Mean = -0.63, 90% CI 2-sided [-1.58 to 0.31], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Test type: Superiority or Other; p = 0.3561, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Mean = -0.52, 90% CI 2-sided [-1.46 to 0.41], Standard Error of Mean 0.57

2. Primary Outcome: Change From Baseline to Month 6 in OMERACT RAMRIS Wrist and MCP Bone Marrow Edema
Description: Bone edema was assessed at 25 anatomic locations: 15 in 1 wrist and 10 in attached hand. Bone edema was defined as a lesion within the trabecular bone, with ill-defined margins and signal characteristics consistent with increased water content. Each bone was scored separately; the scale was 0-3 based on the proportion of bone with edema, as follows 0: no edema; 1: 1-33% of bone edematous; 2: 34-66% of bone edematous; 3: 67-100%. OMERACT RAMRIS total bone edema score for hands/wrists was sum of the individual scores for each location. Thus the maximum score per hand/wrist was 75 (range 0-75). Increasing score=greater severity.
Time Frame: Month 6
Population: Evaluable Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 33 | 29 | 28
score on a scale | -1.26 (0.41) | -1.45 (0.42) | 0.29 (0.42)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Test type: Superiority or Other; p = 0.0089, mixed model repeated measures analysis — 2-sided p-value; alpha= 0.10; Difference in LS Means = -1.55, 90% CI 2-sided [-2.52 to -0.58], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Test type: Superiority or Other; p = 0.0038, mixed model repeated measures analysis — 2-sided p-value; alpha= 0.10; Difference in LS Means = -1.74, 90% CI 2-sided [-2.72 to -0.76], Standard Error of Mean 0.59

3. Secondary Outcome: Change From Baseline to Months 1, 6, and 12 in OMERACT RAMRIS Wrist and MCP Synovitis
Description: as for outcome 1
Time Frame: Months 1, 6, and 12
Population: Evaluable Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 33 | 31 | 35
score on a scale
  Month 1 (n=28,31,35) | -0.42 (0.42) | -0.34 (0.40) | -0.17 (0.38)
  Month 6 (n=33,29,28) | -1.22 (0.40) | -1.29 (0.41) | -0.28 (0.42)
  Month 12 (n=29,26,21) | -2.26 (0.41) | -1.16 (0.43) | -0.66 (0.46)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.6576, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.25, 90% CI 2-sided [-1.19 to 0.69], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.7565, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.17, 90% CI 2-sided [-1.09 to 0.74], Standard Error of Mean 0.55
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.1038, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.94, 90% CI 2-sided [-1.89 to 0.01], Standard Error of Mean 0.58
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0868, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.01, 90% CI 2-sided [-1.98 to -0.04], Standard Error of Mean 0.59
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0103, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.60, 90% CI 2-sided [-2.62 to -0.58], Standard Error of Mean 0.62
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.4350, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.49, 90% CI 2-sided [-1.53 to 0.55], Standard Error of Mean 0.63

4. Secondary Outcome: Change From Baseline to Months 1, 3, and 12 in OMERACT RAMRIS Bone Marrow Edema in Wrist and MCP
Description: Bone edema was assessed at 25 anatomic locations: 15 in 1 wrist and 10 in attached hand. Bone edema was defined as a lesion within the trabecular bone, with ill-defined margins and signal characteristics consistent with increased water content. Each bone was scored separately; the scale was 0â€"3 based on the proportion of bone with edema, as follows 0: no edema; 1: 1â€"33% of bone edematous; 2: 34â€"66% of bone edematous; 3: 67â€"100%. OMERACT RAMRIS total bone edema score for hands/wrists was sum of the individual scores for each location. Thus the maximum score per hand/wrist was 75 (range 0-75). Increasing score=greater severity.
Time Frame: Months 1, 3, and 12
Population: Evaluable Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 30 | 32 | 35
score on a scale
  Month 1 (n=28,31,35) | -0.29 (0.43) | 0.19 (0.41) | 0.11 (0.39)
  Month 3 (n=30,32,31) | -0.77 (0.42) | -0.86 (0.41) | 0.47 (0.41)
  Month 12 (n=29,26,21) | -1.52 (0.42) | -1.70 (0.43) | 0.59 (0.46)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.4890, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.40, 90% CI 2-sided [-1.36 to 0.56], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.8817, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = 0.08, 90% CI 2-sided [-0.85 to 1.02], Standard Error of Mean 0.57
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0351, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.24, 90% CI 2-sided [-2.21 to -0.27], Standard Error of Mean 0.59
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0231, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.32, 90% CI 2-sided [-2.28 to -0.37], Standard Error of Mean 0.58
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0008, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -2.10, 90% CI 2-sided [-3.13 to -1.08], Standard Error of Mean 0.62
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0003, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -2.29, 90% CI 2-sided [-3.32 to -1.25], Standard Error of Mean 0.63

5. Secondary Outcome: Change From Baseline to Months 1, 3, 6, and 12 in OMERACT RAMRIS Wrist and MCP Erosions
Description: Bone erosion assessed at 25 anatomic locations: 15 in 1 wrist and 10 in attached hand. Each site was scored in 1.0 increments from 0 (no damage) to 10 (severe damage), indicating erosion (each unit=10% bone loss) of original articular bone. OMERACT RAMRIS total erosion score for hands/wrists was sum of the individual scores for each location. Thus the maximum score per hand/wrist is 250 (range 0-250). Increasing score=greater severity.
Time Frame: Months 1, 3, 6, and 12
Population: Evaluable Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 33 | 32 | 35
score on a scale
  Month 1 (n=28,31,35) | -0.12 (0.25) | 0.27 (0.25) | 0.27 (0.24)
  Month 3 (n=30,32,31) | -0.12 (0.25) | 0.36 (0.24) | 0.44 (0.25)
  Month 6 (n=33,29,28) | -0.06 (0.25) | -0.02 (0.25) | 0.65 (0.25)
  Month 12 (n=29,26,21) | -0.11 (0.25) | -0.08 (0.25) | 1.18 (0.26)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.2689, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.39, 90% CI 2-sided [-0.96 to 0.19], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.9935, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = 0, 90% CI 2-sided [-0.58 to 0.57], Standard Error of Mean 0.35
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.1086, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.57, 90% CI 2-sided [-1.15 to 0.01], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.8092, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.08, 90% CI 2-sided [-0.66 to 0.49], Standard Error of Mean 0.35
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0463, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.71, 90% CI 2-sided [-1.29 to -0.12], Standard Error of Mean 0.35
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0624, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.67, 90% CI 2-sided [-1.25 to -0.08], Standard Error of Mean 0.35
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0005, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.29, 90% CI 2-sided [-1.90 to -0.69], Standard Error of Mean 0.37
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0008, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.26, 90% CI 2-sided [-1.87 to -0.65], Standard Error of Mean 0.37

6. Secondary Outcome: Modified Total Sharp Score (mTSS) at Months 6 and 12
Description: Modified TSS is a measure of change in joint health. TSS is defined as joint space narrowing score (range 0 [no narrowing] to 168 [high narrowing]) plus (+) erosion score (range is from 0 [no erosion] to 280 [high erosion]). The modified TSS range is from 0 (no damage) to 448 (bad joint status). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Months 6 and 12
Population: Evaluable Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 36 | 37
score on a scale
  Month 6 (n=29,27,28) | 11.28 (0.50) | 10.70 (0.51) | 11.77 (0.52)
  Month 12 (n=26,25,22) | 11.70 (0.51) | 10.69 (0.52) | 12.21 (0.54)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.5019, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.48, 90% CI 2-sided [-1.68 to 0.71], Standard Error of Mean 0.72
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.1462, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.07, 90% CI 2-sided [-2.28 to 0.14], Standard Error of Mean 0.73
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.4900, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.51, 90% CI 2-sided [-1.74 to 0.72], Standard Error of Mean 0.74
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0459, mixed model repeated measures analysis; Difference in LS Means = -1.51, 90% CI 2-sided [-2.76 to -0.27], Standard Error of Mean 0.75

7. Secondary Outcome: Change From Baseline to Months 6 and 12 in mTSS
Description: Modified TSS is a measure of change in joint health. TSS is defined as joint space narrowing score (range 0 [no narrowing] to 168 [high narrowing]) + erosion score (range is from 0 [no erosion] to 280 [high erosion]). The modified TSS range is from 0 (no damage) to 448 (bad joint status). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Months 6 and 12
Population: Evaluable Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 29 | 27 | 28
scores on a scale
  Month 6 (n=29,27,28) | 0.44 (0.50) | -0.14 (0.51) | 0.93 (0.52)
  Month 12 (n=26,25,22) | 0.85 (0.51) | -0.15 (0.52) | 1.36 (0.54)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.5019, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.48, 90% CI 2-sided [-1.68 to 0.71], Standard Error of Mean 0.72
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.1462, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.07, 90% CI 2-sided [-2.28 to 0.14], Standard Error of Mean 0.73
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.4900, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.51, 90% CI 2-sided [-1.74 to 0.72], Standard Error of Mean 0.74
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0459, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.51, 90% CI 2-sided [-2.76 to -0.27], Standard Error of Mean 0.75

8. Secondary Outcome: Joint Space Narrowing (JSN) Scores at Months 6 and 12
Description: JSN score (a component of the modified TSS) is a measure of change in joint health. JSN score range is 0 (no narrowing) to 168 (high narrowing). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Months 6 and 12
Population: Evaluable Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 29 | 27 | 28
score on a scale
  Month 6 (n=29,27,28) | 5.45 (0.34) | 5.11 (0.35) | 5.52 (0.36)
  Month 12 (n=26,25,22) | 5.59 (0.35) | 5.05 (0.36) | 5.88 (0.37)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.8959, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.07, 90% CI 2-sided [-0.89 to 0.76], Standard Error of Mean 0.50
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.4193, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.41, 90% CI 2-sided [-1.25 to 0.43], Standard Error of Mean 0.50
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.5764, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.29, 90% CI 2-sided [-1.13 to 0.56], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.1101, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.83, 90% CI 2-sided [-1.69 to 0.02], Standard Error of Mean 0.52

9. Secondary Outcome: Change From Baseline to Months 6 and 12 in JSN Scores
Description: as for outcome 8
Time Frame: Months 6 and 12
Population: Evaluable Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 29 | 27 | 28
scores on a scale
  Month 6 (n=29,27,28) | 0.29 (0.34) | -0.06 (0.35) | 0.35 (0.36)
  Month 12 (n=26,25,22) | 0.43 (0.35) | -0.12 (0.36) | 0.71 (0.37)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.8959, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.07, 90% CI 2-sided [-0.89 to 0.76], Standard Error of Mean 0.50
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.4193, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.41, 90% CI 2-sided [-1.25 to 0.43], Standard Error of Mean 0.50
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.5764, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.29, 90% CI 2-sided [-1.13 to 0.56], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.1101, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.83, 90% CI 2-sided [-1.69 to 0.02], Standard Error of Mean 0.52

10. Secondary Outcome: Erosion Scores at Months 6 and 12
Description: Erosion score (a component of the modified TSS) is a measure of change in joint health. Erosion score range is from 0 (no erosion) to 280 (high erosion). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Months 6 and 12
Population: Evaluable Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 29 | 27 | 28
scores on a scale
  Month 6 (n=29,27,28) | 5.84 (0.24) | 5.59 (0.25) | 6.26 (0.25)
  Month 12 (n=26,25,22) | 6.10 (0.25) | 5.64 (0.26) | 6.33 (0.27)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.2351, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.42, 90% CI 2-sided [-1.00 to 0.16], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0631, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.67, 90% CI 2-sided [-1.27 to -0.08], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.5369, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.23, 90% CI 2-sided [-0.83 to 0.38], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0620, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.69, 90% CI 2-sided [-1.31 to -0.08], Standard Error of Mean 0.37

11. Secondary Outcome: Change From Baseline to Months 6 and 12 in Erosion Score
Description: as for outcome 10
Time Frame: Months 6 and 12
Population: Evaluable Set; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 29 | 27 | 28
scores on a scale
  Month 6 (n=29,27,28) | 0.16 (0.24) | -0.10 (0.25) | 0.58 (0.25)
  Month 12 (n=26,25,22) | 0.42 (0.25) | -0.05 (0.26) | 0.65 (0.27)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.2351, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.42, 90% CI 2-sided [-1.00 to 0.16], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0631, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.67, 90% CI 2-sided [-1.27 to -0.08], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.5369, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.23, 90% CI 2-sided [-0.83 to 0.38], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0620, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.69, 90% CI 2-sided [-1.31 to -0.08], Standard Error of Mean 0.37

12. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Percent (%) Improvement (ACR20) Response
Description: ACR20 response: greater than or equal to (â‰¥)20% improvement in tender joint count; â‰¥20% improvement in swollen joint count; and â‰¥20% improvement in at least 3 of 5 remaining ACR core measures: Participant's Assessment of Pain; Participant's Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS Non-Responder Imputation (NRI) method: participants with missing values were considered to be non-responders. n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 35 | 36 | 37
percentage of participants
  Month 1 (n=35,35,37) | 42.86 | 57.14 | 29.73
  Month 2 (n=35,36,37) | 68.57 | 61.11 | 40.54
  Month 3 (n=35,36,37) | 77.14 | 61.11 | 48.65
  Month 6 (n=35,36,37) | 74.29 | 66.67 | 45.95
  Month 9 (n=35,36,37) | 71.43 | 58.33 | 43.24
  Month 12 (n=35,36,37) | 71.43 | 61.11 | 43.24
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.2430, Normal approximation to the binomial; Mean Difference (Final Values) = 13.12, 90% CI 2-sided [-5.36 to 31.62], Standard Error of Mean 11.24
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0147, Normal approximation to the binomial; Mean Difference (Final Values) = 27.41, 90% CI 2-sided [8.91 to 45.90], Standard Error of Mean 11.24
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0127, Normal approximation to the binomial; Mean Difference (Final Values) = 28.03, 90% CI 2-sided [9.51 to 46.54], Standard Error of Mean 11.25
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0724, Normal approximation to the binomial; Mean Difference (Final Values) = 20.57, 90% CI 2-sided [1.73 to 39.41], Standard Error of Mean 11.45
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0086, Normal approximation to the binomial; Mean Difference (Final Values) = 28.49, 90% CI 2-sided [10.63 to 46.35], Standard Error of Mean 10.85
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.2808, Normal approximation to the binomial; Mean Difference (Final Values) = 12.46, 90% CI 2-sided [-6.54 to 31.47], Standard Error of Mean 11.55
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0115, Normal approximation to the binomial; Mean Difference (Final Values) = 28.18, 90% CI 2-sided [9.81 to 46.55], Standard Error of Mean 11.16
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.1921, Normal approximation to the binomial; Mean Difference (Final Values) = 15.09, 90% CI 2-sided [-3.94 to 34.12], Standard Error of Mean 11.56
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0115, Normal approximation to the binomial; Mean Difference (Final Values) = 28.18, 90% CI 2-sided [9.81 to 46.55], Standard Error of Mean 11.16
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.1203, Normal approximation to the binomial; Mean Difference (Final Values) = 17.86, 90% CI 2-sided [-1.05 to 36.79], Standard Error of Mean 11.50

13. Secondary Outcome: Percentage of Participants With an ACR 50% Improvement (ACR50) Response
Description: ACR50 response: â‰¥ 50% improvement in tender or swollen joint counts and 50% improvement in 3 of the following 5 criteria: 1) Physician's Global Assessment of Disease Activity, 2) Participant's Assessment of disease activity, 3) Paricipant's Assessment of Pain, 4) Participant's assessment of functional disability via a HAQ, and 5) CRP at each visit.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assess for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 35 | 36 | 37
percentage of participants
  Month 1 (n=35,35,37) | 22.86 | 22.86 | 2.70
  Month 2 (n=35,36,37) | 45.71 | 33.33 | 16.22
  Month 3 (n=35,36,37) | 48.57 | 50.00 | 24.32
  Month 6 (n=35,36,37) | 57.14 | 47.22 | 21.62
  Month 9 (n=35,36,37) | 57.14 | 44.44 | 29.73
  Month 12 (n=35,36,37) | 57.14 | 44.44 | 29.73
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0078, Normal approximation to the binomial; Mean Difference (Final Values) = 20.15, 90% CI 2-sided [7.68 to 32.62], Standard Error of Mean 7.58
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0078, Normal approximation to the binomial; Mean Difference (Final Values) = 20.15, 90% CI 2-sided [7.68 to 32.62], Standard Error of Mean 7.58
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0044, Normal approximation to the binomial; Mean Difference (Final Values) = 29.49, 90% CI 2-sided [12.43 to 46.56], Standard Error of Mean 10.37
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0845, Normal approximation to the binomial; Mean Difference (Final Values) = 17.11, 90% CI 2-sided [0.79 to 33.43], Standard Error of Mean 9.92
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0275, Normal approximation to the binomial; Mean Difference (Final Values) = 24.24, 90% CI 2-sided [6.14 to 42.35], Standard Error of Mean 11.00
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0186, Normal approximation to the binomial; Mean Difference (Final Values) = 25.67, 90% CI 2-sided [7.71 to 43.63], Standard Error of Mean 10.91
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0009, Normal approximation to the binomial; Mean Difference (Final Values) = 35.52, 90% CI 2-sided [17.82 to 53.22], Standard Error of Mean 10.75
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0169, Normal approximation to the binomial; Mean Difference (Final Values) = 25.60, 90% CI 2-sided [7.95 to 43.24], Standard Error of Mean 10.72
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0147, Normal approximation to the binomial; Mean Difference (Final Values) = 27.41, 90% CI 2-sided [8.91 to 45.90], Standard Error of Mean 11.24
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.1882, Normal approximation to the binomial; Mean Difference (Final Values) = 14.71, 90% CI 2-sided [-3.68 to 33.11], Standard Error of Mean 11.18
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0147, Normal approximation to the binomial; Mean Difference (Final Values) = 27.41, 90% CI 2-sided [8.91 to 45.90], Standard Error of Mean 11.24
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.1882, Normal approximation to the binomial; Mean Difference (Final Values) = 14.71, 90% CI 2-sided [-3.68 to 33.11], Standard Error of Mean 11.18

14. Secondary Outcome: Percentage of Participants With an ACR 70% Improvement (ACR70) Response
Description: ACR70 response: â‰¥70% improvement in tender or swollen joint counts and 70% improvement in 3 of the following 5 criteria: 1) Physician's Global Assessment of Disease Activity, 2) Participant's Assessment of Disease Activity, 3) Participant's Assessment of Pain, 4) Participant's Assessment of Functional Disability via a HAQ, and 5) CRP at each visit.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 35 | 36 | 37
percentage of participants
  Month 1 (n=35,35,37) | 8.57 | 2.86 | 0.00
  Month 2 (n=35,36,37) | 31.43 | 22.22 | 5.41
  Month 3 (n=35,36,37) | 25.71 | 27.78 | 10.81
  Month 6 (n=35,36,37) | 34.29 | 30.56 | 21.62
  Month 9 (n=35,36,37) | 31.43 | 33.33 | 18.92
  Month 12 (n=35,36,37) | 22.86 | 33.33 | 21.62
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0700, Normal approximation to the binomial; Mean Difference (Final Values) = 8.57, 90% CI 2-sided [0.78 to 16.35], Standard Error of Mean 4.73
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.3102, Normal approximation to the binomial; Mean Difference (Final Values) = 2.85, 90% CI 2-sided [-1.77 to 7.48], Standard Error of Mean 2.81
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0027, Normal approximation to the binomial; Mean Difference (Final Values) = 26.02, 90% CI 2-sided [11.73 to 40.30], Standard Error of Mean 8.68
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0324, Normal approximation to the binomial; Mean Difference (Final Values) = 16.81, 90% CI 2-sided [3.88 to 29.75], Standard Error of Mean 7.86
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0969, Normal approximation to the binomial; Mean Difference (Final Values) = 14.90, 90% CI 2-sided [0.13 to 29.67], Standard Error of Mean 8.97
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0606, Normal approximation to the binomial; Mean Difference (Final Values) = 16.96, 90% CI 2-sided [2.09 to 31.84], Standard Error of Mean 9.04
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.2276, Normal approximation to the binomial; Mean Difference (Net) = 12.66, 90% CI 2-sided [-4.60 to 29.93], Standard Error of Mean 10.49
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.3827, Normal approximation to the binomial; Mean Difference (Final Values) = 8.93, 90% CI 2-sided [-7.90 to 25.76], Standard Error of Mean 10.23
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.2177, Normal approximation to the binomial; Mean Difference (Final Values) = 12.50, 90% CI 2-sided [-4.18 to 29.20], Standard Error of Mean 10.15
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.1558, Normal approximation to the binomial; Mean Difference (Final Values) = 14.41, 90% CI 2-sided [-2.29 to 31.12], Standard Error of Mean 10.15
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.8997, Normal approximation to the binomial; Mean Difference (Final Values) = 1.23, 90% CI 2-sided [-14.89 to 17.36], Standard Error of Mean 9.80
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.2587, Normal approximation to the binomial; Mean Difference (Final Values) = 11.71, 90% CI 2-sided [-5.34 to 28.76], Standard Error of Mean 10.36

15. Secondary Outcome: Disease Activity Score Based on 28-Joint Count and CRP (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from the swollen joint count and tender joint count using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) less than or equal to (â‰¤)3.2 implied low disease activity and greater than (>)3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) less than (<)2.6 = remission.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, and 12
Population: FAS; n=number of participants assess for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 36 | 36 | 37
score on a scale
  Baseline (n=36,36,37) | 5.14 (0.96) | 5.48 (0.78) | 5.36 (0.80)
  Month 1 (n=33,35,37) | 3.71 (1.15) | 4.03 (0.91) | 4.65 (1.07)
  Month 2 (n=33,33,32) | 2.99 (1.17) | 3.52 (1.15) | 4.21 (1.31)
  Month 3 (n=33,33,31) | 3.06 (1.02) | 3.46 (1.09) | 3.87 (1.43)
  Month 6 (n=31,29,29) | 2.74 (1.15) | 2.75 (0.95) | 3.92 (1.49)
  Month 9 (n=30,28,24) | 2.37 (0.98) | 2.85 (0.90) | 3.58 (1.63)
  Month 12 (n=27,26,20) | 2.49 (1.02) | 2.68 (1.05) | 3.58 (1.40)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -0.22, 90% CI 2-sided [-0.56 to 0.13]
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Baseline; Test type: Superiority or Other; Mean Difference (Final Values) = 0.12, 90% CI 2-sided [-0.19 to 0.43]
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; Mean Difference (Final Values) = -0.94, 90% CI 2-sided [-1.38 to -0.50]
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; Mean Difference (Final Values) = -0.62, 90% CI 2-sided [-1.01 to -0.22]
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; Mean Difference (Final Values) = -1.21, 90% CI 2-sided [-1.73 to -0.70]
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; Mean Difference (Final Values) = -0.69, 90% CI 2-sided [-1.20 to -0.18]
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.81, 90% CI 2-sided [-1.33 to -0.29]
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.41, 90% CI 2-sided [-0.94 to 0.12]
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -1.18, 90% CI 2-sided [-1.75 to -0.61]
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -1.18, 90% CI 2-sided [-1.73 to -0.63]
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; Mean Difference (Final Values) = -1.21, 90% CI 2-sided [-1.81 to -0.61]
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; Mean Difference (Final Values) = -0.73, 90% CI 2-sided [-1.33 to -0.13]
Statistical Analysis 13: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -1.10, 90% CI 2-sided [-1.69 to -0.51]
Statistical Analysis 14: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.90, 90% CI 2-sided [-1.51 to -0.29]

16. Secondary Outcome: Change From Baseline in DAS28-3 (CRP)
Description: DAS28-3 (CRP) was calculated from the swollen joint count and tender joint count using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Tofacitinib (CP-690,550) Plus MTX: Participants received CP-690,550 10 milligrams (mg), tablets, orally (PO), twice daily (BID), and MTX 10 mg per week (mg/week) to 20 mg/week, capsules, PO, for a maximum of 12 months. MTX dose was titrated as follows: 10 mg once weekly for 4 weeks; if well tolerated, then at Month 1 titrate up to 15 mg once weekly for 4 weeks; if well tolerated, then at Month 2 titrate up to 20 mg once weekly for the duration of the study. A single dose reduction of MTX 5 mg was allowed because of lack of tolerance, as long as the participant remained on a dose of at least MTX 10 mg weekly. Participants also received folate supplementation according to local MTX label guidelines and standard of care.
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 33 | 35 | 37
scores on a scale
  Month 1 (n=33,35,37) | -1.61 (0.19) | -1.40 (0.18) | -0.73 (0.18)
  Month 2 (n=33,33,32) | -2.32 (0.19) | -1.88 (0.19) | -1.24 (0.19)
  Month 3 (n=33,33,31) | -2.25 (0.19) | -1.96 (0.19) | -1.57 (0.19)
  Month 6 (n=31,29,29) | -2.54 (0.19) | -2.55 (0.20) | -1.52 (0.19)
  Month 9 (n=30,28,24) | -2.92 (0.20) | -2.43 (0.20) | -1.76 (0.21)
  Month 12 (n=27,26,20) | -2.78 (0.20) | -2.61 (0.20) | -1.77 (0.22)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0010, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.88, 90% CI 2-sided [-1.31 to -0.45], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0102, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.67, 90% CI 2-sided [-1.10 to -0.24], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.08, 90% CI 2-sided [-1.52 to -0.64], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0175, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.64, 90% CI 2-sided [-1.08 to -0.20], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0125, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.68, 90% CI 2-sided [-1.13 to -0.23], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.1457, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.39, 90% CI 2-sided [-0.84 to 0.05], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0003, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.02, 90% CI 2-sided [-1.48 to -0.57], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0002, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.03, 90% CI 2-sided [-1.49 to -0.58], Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.16, 90% CI 2-sided [-1.63 to -0.69], Standard Error of Mean 0.28
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0196, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.67, 90% CI 2-sided [-1.14 to -0.20], Standard Error of Mean 0.28
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0007, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.01, 90% CI 2-sided [-1.50 to -0.52], Standard Error of Mean 0.30
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0049, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.84, 90% CI 2-sided [-1.32 to -0.35], Standard Error of Mean 0.30

17. Secondary Outcome: Disease Activity Score Based on 28-Joint Count and Erythrocyte Sedimentation Rate (DAS28-4 [ESR])
Description: DAS28-4 (ESR) was calculated from swollen joint count and tender joint count using 28 joints count, ESR (millimeters per hour [mm/hour]) and Participant Global Assessment of disease activity (participant rated arthritis activity assessment). Total score range: 0 to 9.4; higher score=more disease activity. DAS28-4 (ESR) â‰¤3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = remission.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, and 12
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 36 | 36 | 37
scores on a scale
  Baseline (n=36,36,37) | 6.25 (0.94) | 6.50 (0.75) | 6.44 (0.78)
  Month 1 (n=34,35,37) | 4.60 (1.37) | 4.93 (1.12) | 5.51 (1.09)
  Month 2 (n=32,33,31) | 3.77 (1.34) | 4.36 (1.40) | 5.05 (1.26)
  Month 3 (n=33,33,31) | 3.66 (1.16) | 4.12 (1.31) | 4.63 (1.63)
  Month 6 (n=30,29,28) | 3.32 (1.45) | 3.51 (1.20) | 4.75 (1.76)
  Month 9 (n=30,28,24) | 3.06 (1.27) | 3.58 (1.10) | 4.17 (1.91)
  Month 12 (n=27,26,20) | 3.02 (1.22) | 3.47 (1.36) | 4.13 (1.76)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -0.19, 90% CI 2-sided [-0.53 to 0.15]
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Baseline; Test type: Superiority or Other; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-0.24 to 0.36]
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; Mean Difference (Final Values) = -0.91, 90% CI 2-sided [-1.40 to -0.42]
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; Mean Difference (Final Values) = -0.58, 90% CI 2-sided [-1.01 to -0.14]
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; Mean Difference (Final Values) = -1.28, 90% CI 2-sided [-1.82 to -0.73]
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; Mean Difference (Final Values) = -0.69, 90% CI 2-sided [-1.25 to -0.13]
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.96, 90% CI 2-sided [-1.55 to -0.38]
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.51, 90% CI 2-sided [-1.12 to 0.11]
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -1.43, 90% CI 2-sided [-2.13 to -0.72]
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; Mean Difference (Final Values) = -1.24, 90% CI 2-sided [-1.91 to -0.57]
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; Mean Difference (Final Values) = -1.11, 90% CI 2-sided [-1.84 to -0.39]
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; Mean Difference (Final Values) = -0.59, 90% CI 2-sided [-1.30 to 0.13]
Statistical Analysis 13: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -1.11, 90% CI 2-sided [-1.84 to -0.39]
Statistical Analysis 14: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.66, 90% CI 2-sided [-1.43 to 0.11]

18. Secondary Outcome: Change From Baseline in DAS28-4 (ESR)
Description: DAS28-4 (ESR) was calculated from swollen joint count and tender joint count using 28 joints count, ESR (millimeters per hour [mm/hour]) and Participant Global Assessment of disease activity (participant rated arthritis activity assessment). Total score range: 0 to 9.4; higher score=more disease activity.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS; n=number of participants assessed for the specified parameter at a given visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 35 | 37
scores on a scale
  Month 1 (n=34,35,37) | -1.77 (0.21) | -1.57 (0.21) | -0.94 (0.20)
  Month 2 (n=32,33,31) | -2.59 (0.22) | -2.08 (0.21) | -1.41 (0.21)
  Month 3 (n=33,33,31) | -2.69 (0.21) | -2.35 (0.21) | -1.80 (0.21)
  Month 6 (n=30,29,28) | -3.02 (0.22) | -2.81 (0.22) | -1.73 (0.22)
  Month 9 (n=30,28,24) | -3.29 (0.22) | -2.72 (0.22) | -2.14 (0.23)
  Month 12 (n=27,26,20) | -3.31 (0.22) | -2.84 (0.22) | -2.18 (0.24)
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0046, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.84, 90% CI 2-sided [-1.32 to -0.35], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0303, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.63, 90% CI 2-sided [-1.11 to -0.15], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0001, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.18, 90% CI 2-sided [-1.69 to -0.68], Standard Error of Mean 0.30
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0255, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.67, 90% CI 2-sided [-1.17 to -0.18], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0035, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.89, 90% CI 2-sided [-1.39 to -0.39], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0683, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.55, 90% CI 2-sided [-1.05 to -0.05], Standard Error of Mean 0.30
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.29, 90% CI 2-sided [-1.81 to -0.78], Standard Error of Mean 0.31
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0006, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.08, 90% CI 2-sided [-1.59 to -0.56], Standard Error of Mean 0.31
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0004, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.15, 90% CI 2-sided [-1.67 to -0.62], Standard Error of Mean 0.32
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0706, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.58, 90% CI 2-sided [-1.10 to -0.05], Standard Error of Mean 0.32
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0008, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -1.13, 90% CI 2-sided [-1.67 to -0.58], Standard Error of Mean 0.33
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0466, mixed model repeated measures analysis — 2-sided p-value; alpha=0.10; Difference in LS Means = -0.66, 90% CI 2-sided [-1.21 to -0.12], Standard Error of Mean 0.33

19. Secondary Outcome: Percentage of Participants With DAS28-3 (CRP) Response (Good or Moderate Improvement)
Description: DAS28-3(CRP) was calculated from the swollen joint count and tender joint count using 28-joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28 categorical responses define a good (absolute: <3.2 or >1.2 improvement from baseline [BL]), moderate (absolute: 3.2-5.1 or 0.6-1.2 change from BL), or no response (absolute: >5.1 or <0.6 change from BL).
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 36 | 37
percentage of participants
  Month 1 (n=33,35,37) | 75.76 | 71.43 | 43.24
  Month 2 (n=34,36,37) | 91.18 | 80.56 | 56.76
  Month 3 (n=34,36,37) | 91.18 | 77.78 | 56.76
  Month 6 (n=34,36,37) | 88.24 | 77.78 | 54.05
  Month 9 (n=34,36,37) | 79.41 | 69.44 | 45.95
  Month 12 (n=34,36,37) | 82.35 | 72.22 | 45.95
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0032, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 32.51, 90% CI 2-sided [14.34 to 50.68], Standard Error of Mean 11.04
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0115, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 28.18, 90% CI 2-sided [9.81 to 46.55], Standard Error of Mean 11.16
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0002, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 34.41, 90% CI 2-sided [18.81 to 50.02], Standard Error of Mean 9.48
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0231, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 23.79, 90% CI 2-sided [6.55 to 41.03], Standard Error of Mean 10.48
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0002, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 34.41, 90% CI 2-sided [18.81 to 50.02], Standard Error of Mean 9.48
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0493, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 21.02, 90% CI 2-sided [3.43 to 38.61], Standard Error of Mean 10.69
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0005, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 34.18, 90% CI 2-sided [17.92 to 50.43], Standard Error of Mean 9.88
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0270, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 23.72, 90% CI 2-sided [6.07 to 41.37], Standard Error of Mean 10.73
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0018, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 33.46, 90% CI 2-sided [15.80 to 51.12], Standard Error of Mean 10.73
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0363, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 23.49, 90% CI 2-sided [5.02 to 41.96], Standard Error of Mean 11.22
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0005, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 36.40, 90% CI 2-sided [19.16 to 53.64], Standard Error of Mean 10.48
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0177, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 26.27, 90% CI 2-sided [8.04 to 44.50], Standard Error of Mean 11.08

20. Secondary Outcome: Percentage of Participants With DAS28-3 (CRP) Score â‰¤3.2
Description: DAS28-3(CRP) was calculated from the swollen joint count and tender joint count using 28-joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3(CRP) â‰¤3.2 implied low disease activity.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 36 | 37
percentage of participants
  Month 1 (n=33,35,37) | 33.33 | 17.14 | 10.81
  Month 2 (n=34,36,37) | 50.00 | 36.11 | 21.62
  Month 3 (n=34,36,37) | 50.00 | 41.67 | 21.62
  Month 6 (n=34,36,37) | 61.76 | 55.56 | 27.03
  Month 9 (n=34,36,37) | 64.71 | 58.33 | 29.33
  Month 12 (n=34,36,37) | 61.76 | 50.00 | 27.03
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0197, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 22.52, 90% CI 2-sided [6.62 to 38.42], Standard Error of Mean 9.66
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.4379, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 6.33, 90% CI 2-sided [-7.09 to 19.76], Standard Error of Mean 8.16
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0093, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 28.37, 90% CI 2-sided [10.40 to 46.34], Standard Error of Mean 10.92
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.1669, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 14.48, 90% CI 2-sided [-2.75 to 31.73], Standard Error of Mean 10.48
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0093, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 28.37, 90% CI 2-sided [10.40 to 46.34], Standard Error of Mean 10.92
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0596, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 20.04, 90% CI 2-sided [2.53 to 37.55], Standard Error of Mean 10.64
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0017, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 34.73, 90% CI 2-sided [16.51 to 52.96], Standard Error of Mean 11.07
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0097, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 28.52, 90% CI 2-sided [10.36 to 46.69], Standard Error of Mean 11.04
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0016, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 34.97, 90% CI 2-sided [16.68 to 53.26], Standard Error of Mean 11.11
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0102, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 28.60, 90% CI 2-sided [10.28 to 46.91], Standard Error of Mean 11.13
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0017, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 34.73, 90% CI 2-sided [16.51 to 52.96], Standard Error of Mean 11.07
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0381, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 22.97, 90% CI 2-sided [4.74 to 41.19], Standard Error of Mean 11.07

21. Secondary Outcome: Percentage of Participants With DAS28-3 (CRP) Score <2.6
Description: DAS28-3(CRP) was calculated from the swollen joint count and tender joint count using 28-joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3(CRP) <2.6 implied remission.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 36 | 37
percentage of participants
  Month 1 (n=33,35,37) | 18.18 | 5.71 | 5.41
  Month 2 (n=34,36,37) | 35.29 | 16.67 | 8.11
  Month 3 (n=34,36,37) | 32.35 | 22.22 | 13.51
  Month 6 (n=34,36,37) | 47.06 | 33.33 | 16.22
  Month 9 (n=34,36,37) | 50.00 | 38.89 | 18.92
  Month 12 (n=34,36,37) | 47.06 | 33.33 | 13.51
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0959, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 12.77, 90% CI 2-sided [0.15 to 25.40], Standard Error of Mean 7.67
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.9544, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 0.30, 90% CI 2-sided [-8.58 to 9.19], Standard Error of Mean 5.40
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0036, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 27.18, 90% CI 2-sided [11.81 to 42.55], Standard Error of Mean 9.34
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.2640, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 8.55, 90% CI 2-sided [-4.04 to 21.16], Standard Error of Mean 7.66
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0544, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 18.83, 90% CI 2-sided [2.72 to 34.95], Standard Error of Mean 9.79
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.3290, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 8.70, 90% CI 2-sided [-5.96 to 23.38], Standard Error of Mean 8.92
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0032, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 30.84, 90% CI 2-sided [13.59 to 48.09], Standard Error of Mean 10.48
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0845, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 17.11, 90% CI 2-sided [0.79 to 33.43], Standard Error of Mean 9.92
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0037, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 31.08, 90% CI 2-sided [13.44 to 48.72], Standard Error of Mean 10.72
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0540, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 19.96, 90% CI 2-sided [2.91 to 37.02], Standard Error of Mean 10.36
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0010, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 33.54, 90% CI 2-sided [16.70 to 50.39], Standard Error of Mean 10.24
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0401, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 19.81, 90% CI 2-sided [3.92 to 35.71], Standard Error of Mean 9.66

22. Secondary Outcome: Percentage of Participants With DAS28-4 (ESR) Response (Good or Moderate Improvement)
Description: DAS28-4(ESR) was calculated from swollen joint count and tender joint count using 28 joints count, ESR (mm/hour) and Participant's Global Assessment of Disease Activity (participant rated arthritis activity assessment). Total score range: 0 to 9.4, higher score=more disease activity. DAS28 categorical responses define a good (absolute: <3.2 or >1.2 improvement from BL), moderate (absolute: 3.2-5.1 or 0.6-1.2 change from BL), or no response (absolute: >5.1 or <0.6 change from BL).
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 35 | 37
percentage of participants
  Month 1 (n=34,35,37) | 67.65 | 62.86 | 29.73
  Month 2 (n=32,33,31) | 85.29 | 69.44 | 59.46
  Month 3 (n=33,33,31) | 91.18 | 69.44 | 51.35
  Month 6 (n=30,29,28) | 85.29 | 77.78 | 51.35
  Month 9 (n=30,28,24) | 82.35 | 72.22 | 45.95
  Month 12 (n=27,26,20) | 79.41 | 69.44 | 45.95
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0005, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 37.91, 90% CI 2-sided [19.83 to 55.99], Standard Error of Mean 10.99
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0028, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 33.12, 90% CI 2-sided [14.87 to 51.38], Standard Error of Mean 11.09
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0105, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 25.83, 90% CI 2-sided [9.21 to 42.45], Standard Error of Mean 10.10
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.3700, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 9.98, 90% CI 2-sided [-8.33 to 28.30], Standard Error of Mean 11.13
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 39.82, 90% CI 2-sided [24.11 to 55.53], Standard Error of Mean 9.54
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.1076, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 18.09, 90% CI 2-sided [-0.40 to 36.59], Standard Error of Mean 11.24
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0008, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 33.94, 90% CI 2-sided [17.13 to 50.75], Standard Error of Mean 10.21
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0139, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 26.42, 90% CI 2-sided [8.74 to 44.10], Standard Error of Mean 10.74
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0005, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 36.40, 90% CI 2-sided [19.16 to 53.64], Standard Error of Mean 10.48
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0177, Normal approximation to the binomial; Mean Difference (Final Values) = 26.27, 90% CI 2-sided [8.04 to 44.50], Standard Error of Mean 11.08
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0018, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 33.46, 90% CI 2-sided [15.80 to 51.12], Standard Error of Mean 10.73
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0363, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 23.49, 90% CI 2-sided [5.02 to 41.96], Standard Error of Mean 11.22

23. Secondary Outcome: Percentage of Participants With DAS28-4 (ESR) â‰¤3.2
Description: DAS28-4(ESR) was calculated from swollen joint count and tender joint count using 28 joints count, ESR (mm/hour) and Participant's Global Assessment of Disease Activity (participant rated arthritis activity assessment). Total score range: 0 to 9.4, higher score=more disease activity. DAS28-4(ESR) â‰¤3.2 implied low disease activity.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 36 | 37
percentage of participants
  Month 1 (n=34,35,37) | 20.59 | 8.57 | 2.70
  Month 2 (n=34,36,37) | 35.29 | 13.89 | 8.11
  Month 3 (n=34,36,37) | 32.35 | 30.56 | 13.51
  Month 6 (n=34,36,37) | 41.18 | 27.78 | 18.92
  Month 9 (n=34,36,37) | 44.12 | 33.33 | 18.92
  Month 12 (n=34,36,37) | 50.00 | 30.56 | 16.22
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.0160, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 17.88, 90% CI 2-sided [5.66 to 30.10], Standard Error of Mean 7.42
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.2798, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 5.86, 90% CI 2-sided [-3.06 to 14.80], Standard Error of Mean 5.43
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.0036, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 27.18, 90% CI 2-sided [11.81 to 42.55], Standard Error of Mean 9.34
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.4287, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 5.78, 90% CI 2-sided [-6.23 to 17.79], Standard Error of Mean 7.30
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0544, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 18.83, 90% CI 2-sided [2.72 to 34.95], Standard Error of Mean 9.79
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0732, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 17.04, 90% CI 2-sided [1.39 to 32.69], Standard Error of Mean 9.51
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0360, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 22.25, 90% CI 2-sided [4.79 to 39.72], Standard Error of Mean 10.61
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.3688, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 8.85, 90% CI 2-sided [-7.35 to 25.07], Standard Error of Mean 9.85
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0182, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 25.19, 90% CI 2-sided [7.63 to 42.76], Standard Error of Mean 10.67
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.1558, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 14.41, 90% CI 2-sided [-2.29 to 31.12], Standard Error of Mean 10.15
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0012, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 33.78, 90% CI 2-sided [16.51 to 51.05], Standard Error of Mean 10.49
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.1426, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Net) = 14.33, 90% CI 2-sided [-1.74 to 30.42], Standard Error of Mean 9.78

24. Secondary Outcome: Percentage of Participants With DAS28-4 (ESR) <2.6
Description: DAS28-4(ESR) was calculated from swollen joint count and tender joint count using 28 joints count, ESR (mm/hour) and Participant's Global Assessment of Disease Activity (participant rated arthritis activity assessment). Total score range: 0 to 9.4, higher score=more disease activity. DAS28-4(ESR) <2.6 implied remission.
Time Frame: Months 1, 2, 3, 6, 9, and 12
Population: FAS NRI; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Number analyzed (Participants) | 34 | 36 | 37
percentage of participants
  Month 1 (n=34,35,37) | 5.88 | 2.86 | 0.00
  Month 2 (n=34,36,37) | 17.65 | 5.56 | 2.70
  Month 3 (n=34,36,37) | 23.53 | 2.78 | 13.51
  Month 6 (n=34,36,37) | 29.41 | 13.89 | 13.51
  Month 9 (n=34,36,37) | 35.29 | 13.89 | 16.22
  Month 12 (n=34,36,37) | 32.35 | 19.44 | 13.51
Statistical Analysis 1: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.1449, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 5.88, 90% CI 2-sided [-0.75 to 12.52], Standard Error of Mean 4.03
Statistical Analysis 2: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 1; Test type: Superiority or Other; p = 0.3102, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 2.85, 90% CI 2-sided [-1.77 to 7.48], Standard Error of Mean 2.81
Statistical Analysis 3: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Tofacitinib (CP-690,550); Month 2; Test type: Superiority or Other; p = 0.0342, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 14.94, 90% CI 2-sided [3.32 to 26.55], Standard Error of Mean 7.06
Statistical Analysis 4: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 2; Test type: Superiority or Other; p = 0.5400, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 2.85, 90% CI 2-sided [-4.80 to 10.51], Standard Error of Mean 4.65
Statistical Analysis 5: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.2759, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 10.01, 90% CI 2-sided [-5.10 to 25.13], Standard Error of Mean 9.19
Statistical Analysis 6: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 3; Test type: Superiority or Other; p = 0.0859, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = -10.73, 90% CI 2-sided [-21.02 to -0.45], Standard Error of Mean 6.25
Statistical Analysis 7: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.0985, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 15.89, 90% CI 2-sided [0.06 to 31.73], Standard Error of Mean 9.62
Statistical Analysis 8: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 6; Test type: Superiority or Other; p = 0.9628, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 0.37, 90% CI 2-sided [-12.86 to 13.61], Standard Error of Mean 8.05
Statistical Analysis 9: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.0612, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 19.07, 90% CI 2-sided [2.31 to 35.84], Standard Error of Mean 10.19
Statistical Analysis 10: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 9; Test type: Superiority or Other; p = 0.7807, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = -2.32, 90% CI 2-sided [-16.08 to 11.43], Standard Error of Mean 8.36
Statistical Analysis 11: Comparison: Tofacitinib (CP-690,550) Plus MTX vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.0544, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 18.83, 90% CI 2-sided [2.72 to 34.95], Standard Error of Mean 9.79
Statistical Analysis 12: Comparison: Tofacitinib (CP-690,550) vs Methotrexate; Month 12; Test type: Superiority or Other; p = 0.4937, Normal approximation to the binomial — 2-sided p-value; alpha=0.10; Mean Difference (Final Values) = 5.93, 90% CI 2-sided [-8.32 to 20.18], Standard Error of Mean 8.66

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 28 calendar days after the last administration of investigational product.
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tofacitinib (CP-690,550) Plus MTX | Tofacitinib (CP-690,550) | Methotrexate
Serious Adverse Events (participants affected / at risk) | 2/36 | 1/36 | 2/37
Other Adverse Events (participants affected / at risk) | 24/36 | 31/36 | 29/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (CP-690,550) Plus MTX (N=36) | Tofacitinib (CP-690,550) (N=36) | Methotrexate (N=37)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib (CP-690,550) Plus MTX (N=36) | Tofacitinib (CP-690,550) (N=36) | Methotrexate (N=37)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 1 (1) | 2 (2)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (6) | 0 (0) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 5 (5)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine fibrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No